CLINICAL TRIAL: NCT06791161
Title: A Multicenter Prospective Cohort Study of Adjuvant Therapy for BRCA1/2 Mutated Hormone Receptor-positive HER2-negative Early High-risk Breast Cancer
Status: Enrolling by invitation | Type: Observational
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, PENG YUAN, Head of department, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Other Study IDs: NCC5094
Record Dates: First submitted 2025-01-17; First posted 2025-01-24 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-01

CONDITIONS: Breast
Keywords: BRCA1/2 mutation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (1):
- BRCA1/2 mutated HR+HER2- early high-risk breast cancer
  Interventions: Drug: Endocrine drug +CDK4/6 inhibitor or PRAP inhibitor or Endocrine drug +CDK4/6 inhibitor+PARP inhibitor

INTERVENTIONS:
Drug: Endocrine drug +CDK4/6 inhibitor or PRAP inhibitor or Endocrine drug +CDK4/6 inhibitor+PARP inhibitor — BRCA1/2 mutated hormone receptor-positive HER2-negative early high-risk breast cancer is treated with 3 3 treatment options after surgery：Endocrine drug +CDK4/6 inhibitor or PRAP inhibitor or Endocrine drug +CDK4/6 inhibitor+PARP inhibitor

SUMMARY:
To evaluate the efficacy and safety of different adjuvant treatment options after surgery for early high-risk breast cancer with BRCA1/2 mutation HR+/HER2

ELIGIBILITY:
Inclusion Criteria:

* ECOG score 0-1
* ER>10%, PR>10%, HER2(0)/HER2(1+)/HER2(2+) and no amplification of FISH
* BRCA1/2 gene mutation
* No other site metastases were detected by imaging evaluation after surgical treatment
* Non-PCR breast cancer after neoadjuvant therapy, or breast cancer with postoperative pathology indicating ≥pN2
* The patient had no major organ dysfunction

Exclusion Criteria:

* Allergic to the investigational drug, inability to take the drug orally, or refusal of the medication regimen
* Has been enrolled in another study or has been discontinued for less than or equal to 4 weeks
* There is serious dysfunction of vital organs (heart, liver, kidney)
* Patients with other malignancies, except cured non-melanoma skin cancer, cervical carcinoma in situ and other tumors that have been cured for at least 5 years
* In other acute infectious disease or chronic infectious disease activity period
* A history of uncontrolled seizures, central nervous system disorders, or mental disorders
* There is a known history of human immunodeficiency virus

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: BRCA gene mutation HR+/HER2- Early high-risk breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-01-19 (Actual); Primary Completion 2030-01-18 (Estimated); Study Completion 2035-01-18 (Estimated)

PRIMARY OUTCOMES:
Invasive Disease-Free Survival rate | 3 years

SECONDARY OUTCOMES:
Distant relapse-free survival rate | 3 years
Overall survival rate | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No